CLINICAL TRIAL: NCT02314364
Title: A Phase II Trial of Integrating Stereotactic Body Radiation Therapy With Selective Targeted Therapy in Stage IV Oncogene-driven Non-Small Cell Lung Cancer
Brief Title: A Trial of Integrating SBRT With Targeted Therapy in Stage IV Oncogene-driven NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Henning Willers, M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-370
Record Dates: First submitted 2014-11-20; First posted 2014-12-11 (Estimated); Results first posted 2024-03-04 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer Metastatic; Targetable Oncogenes (EGFR, ALK, ROS1)
Keywords: Non-small cell lung cancer; Metastatic; EGFR; ALK; ROS1; Stereotactic Body Radiation Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — Radiosurgery; Protons; Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic body radiation therapy (SBRT) with protons or photons (Experimental): * SBRT dosage determined by treating physician
  * Patients will continue to receive standard of care (SOC) tyrosine kinase inhibitors (TKI) in the intervals between SBRT courses, as well as after the completion of SBRT
  * If there is more than one active site of cancer, additional site(s) will be treated with stereotactic treatment courses. The total duration of SBRT courses (from the first day of any SBRT course to the last day of any SBRT course) will not exceed 4 months.
  Interventions: Radiation: SBRT with protons or photons

INTERVENTIONS:
Radiation: SBRT with protons or photons
  Other Names: Stereotactic body radiation therapy

SUMMARY:
This research study is studying a type of radiation therapy called Stereotactic Body Radiation Therapy (SBRT) as a possible treatment for stage IV non-small cell lung cancer (NSCLC) that has a mutated epidermal growth factor receptor (EGFR) or or displaced anaplastic lymphoma receptor tyrosine kinase (ALK) or ROS proto-oncogene 1 (ROS1) gene (= oncogene-driven NSCLC) and for which the subject has been receiving treatment with a targeted biological agent such as erlotinib, crizotinib, or other drugs.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. The investigational intervention in this study is SBRT with proton or photon radiation (explained below). "Investigational" means that the intervention is being studied. SBRT and proton radiation therapy are FDA approved radiation delivery systems. However, using it as a treatment for stage IV NSCLC is still investigational.

SBRT is a specialized, technologically advanced type of external beam radiation therapy that pinpoints high doses of radiation directly on the cancer. Because of high precision, these treatments spare healthy tissue and are associated with fewer side effects. SBRT is very different from conventional therapy where radiation is delivered in small doses given daily over the course of several weeks. For SBRT, the total dose of radiation is typically administered in 4-5 daily sessions. SBRT can be delivered with standard, so called photon radiation, or proton beam. Neither of these two types of radiation is generally superior over the other. There are technical differences between these two, and depending on tumor location, size, shape, and other factors, the investigators will decide which type of radiation to use for which treatment.

After the screening procedures confirm you are eligible to participate in the research study:

- Each participant will receive stereotactic treatment course (SBRT with protons or photons) to the area of their tumor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) with any actionable mutation or translocation in EGFR, ALK, or ROS1
* Stage IV disease (AJCC Staging system 7th edition)
* Within 6 months of initiating their first TKI treatment regimen
* Stable or responding systemic disease to TKI (no evidence of progression) on the most recent staging studies. The complete extent of the current residual systemic disease must be deemed amenable to SBRT as per review of imaging studies by a radiation oncologist, based on the following criteria:

  * Lung: 1-3 lesions (including the primary) of maximum size 5 cm in longest diameter. A minimum size 1 cm in the longest diameter is recommended. (Patients with a malignant pleural effusion prior to the start of TKI therapy will be considered eligible for SBRT if there is complete radiographic resolution of the effusion while on systemic therapy);
  * Spine: Bone lesions must be limited to the spine. A maximum of 2 spinal metastases will be considered for SBRT, with each site spanning 1-3 vertebral bodies. A minimum size of 1 cm in longest diameter is recommended. SBRT may target sclerotic lesions that persist following TKI therapy;
  * GI: 1-4 liver metastases of maximum size 5 cm in longest diameter and/or 1-2 adrenal metastases of maximum 4 cm size in longest diameter. A minimum size of 1 cm in longest diameter is recommended.

In addition:

* CNS: 1-4 brain metastases of maximum size 3cm in longest diameter. However, these should be treated with standard-of-care SRS and will not be defined as target lesions for purposes of this protocol.
* A maximum number of 5 target lesions outside the brain, excluding the lung primary, is recommended to ensure that enrollment is limited to patients with low-burden disease and that treatments can be delivered within the specified time frame.

  * History of prior radiation therapy to brain or skeleton is allowed, but should have occurred > 2 months from enrollment.
  * Age at least 18 years.
  * Life expectancy of greater than 6 months.
  * ECOG performance status ≤ 2.
  * Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A negative serum or urine pregnancy test within 2 weeks of registration for women of childbearing potential is required.
  * Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Residual hilar or mediastinal lymph node disease (size > 1cm in short-axis diameter on CT). Non-malignant etiologies for enlarged lymph nodes may be evaluated per standard clinical practice.
* Participants who have received prior radiation therapy to anatomical sites other than brain or skeleton.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who are pacemaker or defibrillator-dependent as these devices may not be operated concurrently with delivery of proton beam radiation.
* Pregnant or lactating women, as treatment involves unforeseeable risks to the embryo or fetus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-12; Primary Completion 2021-11-10 (Actual); Study Completion 2023-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henning Willers, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stereotactic body radiation therapy (SBRT) with protons or photons
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Stereotactic Body Radiation Therapy (SBRT) With Protons or Photons
Number analyzed (Participants) | 27
Age, Continuous [Median (Full Range); unit: years] | 59 [42 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: 1-year Frequency of Distant Failures (DF) After Stereotactic Body Radiation Therapy (SBRT)
Description: Distant failures (DF) are defined as metastases outside areas that originally contained disease. The 1-year frequency of DF is defined as the percentage of patients that experienced a DF, respectively, over the course of one year.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stereotactic body radiation therapy (SBRT) with protons or photons
Number analyzed (Participants) | 27
percentage of participants | 19 [7 to 36]

2. Secondary Outcome: Percentage of Participants With Grade 3 or Higher Toxicities Related to Stereotactic Body Radiation Therapy (SBRT)
Description: Adverse events were graded according to Common Terminology Criteria for Adverse Events (CTCAE v4.0). Treatment-related toxicities are defined as adverse events assessed as related to SBRT.
Time Frame: Up to 8.4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic body radiation therapy (SBRT) with protons or photons
Number analyzed (Participants) | 27
Participants | 0

3. Secondary Outcome: Median Progression Free Survival
Description: Progression free survival is defined as the duration of time from the start of standard of care TKI (tyrosine kinase inhibitor) therapy until objective progressive disease or death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 7.65 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stereotactic body radiation therapy (SBRT) with protons or photons
Number analyzed (Participants) | 27
months | 23.4 [14 to 53]

4. Secondary Outcome: Median Overall Survival
Description: Overall survival is defined as the duration of time from the start of documented tyrosine kinase inhibitor (TKI) therapy to the time of death.
Time Frame: Up to 8.4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stereotactic body radiation therapy (SBRT) with protons or photons
Number analyzed (Participants) | 27
months | 59.6 [42.3 to NA] — Too few events occurred to estimate the upper confidence limit for median overall survival.

5. Secondary Outcome: 2-year Overall Survival
Description: Overall survival is defined as the duration of time from the start of documented tyrosine kinase inhibitor (TKI) therapy to the time of death. The 2-year overall survival is defined as the percentage of participants who were alive 2 years after the start of documented tyrosine kinase inhibitor (TKI) therapy.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stereotactic body radiation therapy (SBRT) with protons or photons
Number analyzed (Participants) | 27
percentage of participants | 88 [68 to 96]

6. Secondary Outcome: 2-year Local Failure (LF) of Lesions Treated With Stereotactic Body Radiation Therapy (SBRT)
Description: Local failure is defined as progressive disease in target lesions treated with SBRT. The 2-year LF rate is the percentage of participants who experienced local failure within 2 years of completing SBRT.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stereotactic body radiation therapy (SBRT) with protons or photons
Number analyzed (Participants) | 27
percentage of participants | 11 [3 to 27]

ADVERSE EVENTS:
Time Frame: Up to 8.4 years
Arm/Group | Stereotactic body radiation therapy (SBRT) with protons or photons
All-Cause Mortality (participants affected / at risk) | 12/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 27/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stereotactic body radiation therapy (SBRT) with protons or photons (N=27)
Abdominal Distension (Gastrointestinal disorders) | 3
Abdominal Pain (Gastrointestinal disorders) | 3
Abducens nerve disorder (Nervous system disorders) | 1
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 5
Amnesia (Nervous system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 3
Anxiety (Psychiatric disorders) | 4
Apnea (Respiratory, thoracic and mediastinal disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Aspartate aminotransferase increased (Investigations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 11
Blood bilirubin increased (Investigations) | 2
Blurred vision (Eye disorders) | 4
Bruising (Injury, poisoning and procedural complications) | 2
Cataract (Eye disorders) | 3
Chest pain - cardiac (Cardiac disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 4
Chills (General disorders) | 5
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1
Confusion (Psychiatric disorders) | 3
Conjunctivitis (Eye disorders) | 2
Constipation (Gastrointestinal disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Dehydration (Metabolism and nutrition disorders) | 2
Depression (Psychiatric disorders) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 2
Diarrhea (Gastrointestinal disorders) | 19
Dizziness (Nervous system disorders) | 7
Dry eye (Eye disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 12
Dysgeusia (Nervous system disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 3
Dysphasia (Nervous system disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12
Ear pain (Ear and labyrinth disorders) | 1
Edema face (General disorders) | 1
Edema limbs (General disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Esophageal pain (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 2
Alternating exophoria (Eye disorders) | 1
Dysconjugate gaze (Eye disorders) | 1
Eyelid function disorder (Eye disorders) | 1
Fall (Injury, poisoning and procedural complications) | 5
Fatigue (General disorders) | 16
Fecal incontinence (Gastrointestinal disorders) | 1
Fever (General disorders) | 4
Flashing lights (Eye disorders) | 1
Flu like symptoms (General disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Gait disturbance (General disorders) | 7
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 9
Hearing impaired (Ear and labyrinth disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Hepatitis viral (Infections and infestations) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hot flashes (Vascular disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypersomnia (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hypotension (Vascular disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Insomnia (Psychiatric disorders) | 7
Increased neutrophils (Investigations) | 1
Laryngitis (Infections and infestations) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Lipase increased (Investigations) | 1
Localized edema (General disorders) | 2
Lymph gland infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 12
Malaise (General disorders) | 2
Memory impairment (Nervous system disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1
Leg cramps (Musculoskeletal and connective tissue disorders) | 1
Lower left extremity numbness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 12
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 3
Non-cardiac chest pain (General disorders) | 5
Oculomotor nerve disorder (Nervous system disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain (General disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Palpitations (Cardiac disorders) | 3
Papulopustular rash (Infections and infestations) | 1
Paresthesia (Nervous system disorders) | 3
Paronychia (Infections and infestations) | 7
Pelvic pain (Reproductive system and breast disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1
Platelet count decreased (Investigations) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6
Presyncope (Nervous system disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 9
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Rash pustular (Infections and infestations) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Rectal perforation (Gastrointestinal disorders) | 1
neurogenic sensory cystopathy (Renal and urinary disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis infective (Infections and infestations) | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Seizure (Nervous system disorders) | 1
Serum amylase increased (Investigations) | 1
Serum sickness (Immune system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Sinusitis (Infections and infestations) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin infection (Infections and infestations) | 2
Dermatoheliosis (Skin and subcutaneous tissue disorders) | 1
Cracking of fingernails (Skin and subcutaneous tissue disorders) | 1
Soft tissue infection (Infections and infestations) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Transient ischemic attacks (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Upper respiratory infection (Infections and infestations) | 3
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Urinary tract infection (Infections and infestations) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Watering eyes (Eye disorders) | 2
Weight gain (Investigations) | 2
Weight loss (Investigations) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
White blood cell decreased (Investigations) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/64/NCT02314364/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT02314364/ICF_001.pdf